CLINICAL TRIAL: NCT02550171
Title: The BioGene Bank Cohort Study is a Collection of Human Blood Samples (DNA and Plasma) Along With De-identified (Coded) Health Information, Questionnaire Responses on Environment and History of Family Disease to be Used for Research
Brief Title: BioGene Bank Cohort Study for Approved Research Requests
Acronym: BGB
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Peter Gregersen, Center Head: Robert S. Boas Center for Genomics and Human Genetics, Northwell Health
Other Study IDs: 08-094; Other (Other: North Shore Long Island Jewish Health System)
Record Dates: First submitted 2013-10-09; First posted 2015-09-15 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Healthy; Chronic Disease
Keywords: Biobank; Genetics; DNA; Cohort; normal control
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The BioGene bank: Is a centralized collection of human blood samples along with de-identified (coded) health information, environmental factors, family disease histories and information from DNA. Limited to the NSLIJHS catchment area.

DETAILED DESCRIPTION:
The purpose of the BioGene Bank Cohort is to collect blood and store DNA from blood, along with health information to study how genetic variation in the population is associated with particular diseases, treatments and medical outcomes. Investigators may study the entire range of diseases and medical problems that exist within the NSLIJHS, including medical, surgical, psychiatric, pediatric and obstetric conditions. The specimens and medical information will be kept at a central Biorepository. This research study does not involve any treatment and individual research results are not provided.

ELIGIBILITY:
Inclusion Criteria:

* Anyone receiving care at the NS LIJ Health System would be eligible to join the BioGene Bank Cohort.
* Participants' family members who may or may not have medical records at NSLIJHS.

Exclusion Criteria:

* Patients unable to give consent because they are decisionally impaired or have a language barrier that cannot be overcome.
* Patients unable to provide a blood sample because it would adversely affect their health or who refuse to provide blood sample or share future discarded biological samples.
* Patients <10kg in weight

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anyone receiving care at the NS LIJ Health System and family members.
Sampling Method: Non-Probability Sample
Enrollment: 7056 (Actual)
Dates: Start 2009-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time from symptoms to diagnosis of autoimmune diseases | 10 years
  Documentation of symptoms to diagnosis of autoimmune disease(s)

SECONDARY OUTCOMES:
Chart Review of Participants who are diagnosed with autoimmune disease | average of 10 years
  Review of electronic health records with genetic data to possibly predict development of autoimmune disease

CONTACTS AND LOCATIONS:
Overall Officials: Peter K Gregersen, MD, Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No